CLINICAL TRIAL: NCT03310710
Title: Heparin Bonded Balloon-expandable Stent Grafts for Branches of a Fenestrated Endovascular Aortic Repair Graft
Brief Title: VIABAHN BX Used in Fenestrated EVAR Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Kongteng Tan, Principal Investigator, University Health Network, Toronto
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAPCR 16-5084
Record Dates: First submitted 2017-10-05; First posted 2017-10-16 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Aortic Aneurysm, Abdominal
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Intervention Model Description: Treatment with Viabahn BX stents
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment with Viabahn BX stent (Experimental): Treatment with Viabahn BX stent as branch device in fenestrated EVAR
  Interventions: Device: Viabahn BX stent

INTERVENTIONS:
Device: Viabahn BX stent — Viabahn BX stent graft used as the branch device with a fenestrated EVAR graft

SUMMARY:
Fenestrated endovascular abdominal aortic aneurysm repair (FEVAR) is a procedure to treat abdominal aortic aneurysms which are not amenable to conventional repair or stenting. A stent is placed in the aorta and confines blood flow to a normal diameter lumen to remove pressure on the diseased aortic wall. Fenestrations (custom holes in the graft) are necessary to maintain blood flow to abdominal organs when the aneurysm sac extends to far proximally. These fenestrations are then typically aligned with their respective vessels using covered stents. These stents also help keep the arteries open.

Unfortunately some of the stents currently used occlude either immediately or over time, which can lead to organ failure, morbidity and death. A recent advancement in stent design has heparin bonded to the stent surface which prevents clot from forming. This new design has been shown to help maintain stent patency in other parts of the body. The investigators believe it may do the same for FEVAR patients. The proposed study is a 20-patient pilot to assess the safety of substituting a heparin bonded stent graft for FEVAR branches over a period of one year. Patients who are deemed eligible for FEVAR by a UHN multidisciplinary vascular conference will be recruited to the study. All the branches in their FEVAR will use the Viabahn BX stent in place of the current standard of care stent. They will then be followed per the standard of care for one year. Adverse events will be recorded and the rate of occlusion will be assessed based on CT imaging.

The investigators hypothesize that using heparin bonded stent grafts is safe and they will have a low rate of occlusion.

DETAILED DESCRIPTION:
FEVAR branches can occlude jeopardizing perfusion of the organs they supply. A recent study has shown the rate of patency as 95.7% at 1 year and 88.6% at 4 years. Pooled analysis has shown a 4.5% rate of renal artery occlusion during 12 month follow up with 2.3% going on to dialysis and 1.4% requiring permanent dialysis. 1.8% of patients can go on to have mesenteric stenosis though these have been due to technical issues with the stents.

Studies have previously shown that the patency of vascular grafts can be improved by bonding heparin bonding to the surface of a graft material. For example in surgical bypass a Dacron graft bonded with heparin outperformed a conventional PTFE graft in terms of patency and clinical outcomes. Endovascular stent grafting with heparin bonded PTFE has also been shown to be superior to PTFE alone with a primary patency of 86.4% vs 79.9% in femoropopliteal disease. A recent trial has demonstrated impressive patency of 73% in long segment femoropopliteal disease (TASC C and D lesions) using a self expanding version of the heparin bonded, covered, Viabahn stent graft. Heparin bonded stent grafts have shown promise in preserving patency of other vessels. A pilot study demonstrating the safety of using the Viabahn Bx in FEVAR will support the rationale for larger studies of this question including randomization between conventional and heparin bonded stent grafts.

ELIGIBILITY:
Inclusion Criteria:

* Fenestrated EVAR candidates as determined by the vascular interdisciplinary conference at UHN

Exclusion Criteria:

* Unable to provide informed consent (legally authorized representative is acceptable)
* Age < 18
* Patients with a known hypersensitivity to heparin, including those patients who have had a previous incidence of HIT (heparin induced thrombocytopenia) type II.
* Currently participating in another investigative clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-02-13 (Actual); Primary Completion 2018-10-17 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
Technical success related the Viabahn BX stent graft when used as the branch device with a fenestrated EVAR graft. | Intraoperative (End of EVAR surgery)
  Successful deployment of the Viabahn BX stent graft without major adverse events, such as occlusion of the arteries, at the end of the fenestrated EVAR surgery.
Adverse event related to the Viabahn BX stent graft when used as the branch device with a fenestrated EVAR graft. | 12 months post surgery
  Any stent related adverse event, such as occlusion of the stent and stent fracture

CONTACTS AND LOCATIONS:
Overall Officials: Kong Teng Tan, MD, Principal Investigator — University Health Network, Toronto General Hospital
Locations (1):
- University Health Network, Toronto General Hospital, Toronto, Ontario, Canada